CLINICAL TRIAL: NCT07006766
Title: Bucatini Pasta, Japanese Shirataki Konjac Noodles, and Artificial Vessels: In Search of the Ideal Low-cost Vessel Simulator for Microsurgical Education
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-1534; A539730 (Other: UW Madison)
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Surgical Procedure, Unspecified
Keywords: microsuture; microsurgery; surgical training; microsurgical education; global; accessibility; noodle; synthetic; vessel; anastomosis; patency; education; outreach; low-cost; microsurgical simulation; simulation; vessel simulator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Microsurgical training: Participants will complete pre-exercise surveys, attempt 4 microsurgical anastomoses, and complete post-exercise surveys.
  Interventions: Other: Microsurgical Training Models

INTERVENTIONS:
Other: Microsurgical Training Models — Four models will be compared: Japanese shirataki konjac noodle, "Dragon skin" silicone vessel, standard silicone vessel from Microsurgery and Regenerative Medicine (MSRM) lab, and the "blue-blood" chicken thigh model.

SUMMARY:
The aim of this study is to assess the strengths and weaknesses of training models that are accessible, reproducible, and geared toward new learners. Specifically, the investigators aim to compare the four following models: Japanese shirataki konjac noodle, "Dragon skin" silicone vessel, standard silicone vessel, and the "blue-blood" chicken thigh model. This information will be valuable in assessing the utility of implementing a Japanese shirataki konjac noodle model in beginner microsurgical courses for both local and global education and outreach.

DETAILED DESCRIPTION:
The significant benefit Japanese shirataki konjac noodle as a model for microsurgical simulation training is that they are very cost effective and allow for acquisition of microsurgical skills in a low stake environment. This is particularly useful for the microsurgery novice to become familiar with the tools and basics of placing microsuture.

In this study, the evaluator will complete a "pre-exercise" survey online using a laptop in the microsurgical work space. The evaluator will be oriented to the work space and then attempt to perform an end-to-end anastomoses on each of the four models.

The following three measurements will be taken: time to perform anastomosis, number of stitches, and patency (Yes/No).

Following these trials, the evaluator will take a "post-exercise" survey. This survey will obtain the evaluator's assessment of the models including most and least valuable aspects of each model, ease & comfort of placing a suture, and microsuture/microsurgical tool handling. Only one evaluator will be in the microsurgical lab space at one time. All study tasks will take approximately 1-2 hours. The individuals with no formal surgery/microsurgery education will be guided by an expert microsurgeon throughout the anastomoses. No varying instructional techniques will be assessed; all participants without formal training will receive identical guidance from the expert microsurgeon. The surgical residents will not need supervision or guidance. The training surgeries will not be offered if people are unable to take the research surveys.

ELIGIBILITY:
Inclusion Criteria:

* Participant is able to commit 1-2 hours to the study.
* Participants must either be a surgical resident or an individual with no formal surgery/microsurgery education. Five participants will be placed into each of these two categories.

Exclusion Criteria:

* Participant is unable to commit 1-2 hours to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgical residents or individual with no formal microsurgical education.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-12-23 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Time to Perform Anastomosis | up to 30 min
Number of Stitches | up to 30 min
Patency (either Yes or No) | up to 30 min
  Patency is the condition of being 'open'.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Poore, MD, PhD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- UW School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prunieres GJ, Taleb C, Hendriks S, Miyamoto H, Kuroshima N, Liverneaux PA, Facca S. Use of the Konnyaku Shirataki noodle as a low fidelity simulation training model for microvascular surgery in the operating theatre. Chir Main. 2014 Apr;33(2):106-11. doi: 10.1016/j.main.2013.12.003. Epub 2014 Feb 4. PMID 24603055
- [Background] Mohammad S, Hanstein R, Lo Y, Levy IM. Validating a Low-Fidelity Model for Microsurgical Anastomosis Training. JB JS Open Access. 2021 Jul 16;6(3):e20.00148. doi: 10.2106/JBJS.OA.20.00148. eCollection 2021 Jul-Sep. PMID 34291182
- [Background] Ng ZY, Honeyman C, Lellouch AG, Pandya A, Papavasiliou T. Smartphone-Based DIY Home Microsurgical Training with 3D Printed Microvascular Clamps and Japanese Noodles. Eur Surg Res. 2023;64(2):301-303. doi: 10.1159/000521439. Epub 2021 Dec 15. PMID 34915484